CLINICAL TRIAL: NCT03971396
Title: The Chest Physiotherapy and Breathing Exercises Management of Patients Following Open Heart Surgery: a National Survey of Practice in Turkey.
Status: Completed | Type: Observational
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Collaborators: Koşuyolu Kartal Heart Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Halime Sinem Barutçu, Physiotherapist, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Other Study IDs: DrLutfiKirdarTRH
Record Dates: First submitted 2019-05-30; First posted 2019-06-03 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Chest Physiotherapy
Keywords: open cardiac surgery; breathing exercises; chest physiotherapy
MeSH Terms: interventions — Critical Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Physiotherapists working in intensive care — Physiotherapists working in intensive care will be reached by mail or telephone. Physiotherapists will be asked to complete the prepared questionnaire.

SUMMARY:
Chest physiotherapy and breathing exercises are an important non-pharmacological treatment modality in order to prevent and minimize postoperative respiratory complications in patients undergoing open heart surgery. Different respiratory techniques are used after cardiac surgery, but there is no opinion about which technique or exercise is effective. The purpose of this study, practical application of chest physiotherapy to patients who have had open heart surgery in Turkey and to identify methods of breathing exercises.

DETAILED DESCRIPTION:
In this study, cardiovascular surgery in Turkey to employees or physiotherapist who worked in intensive care units was planned as e-mail or by reaching to answer the survey questions via telephone.

The universe of study in Turkey cardiovascular surgery physiotherapists are all actively working or have worked in intensive care.

ELIGIBILITY:
Inclusion Criteria:

* To worked or still working in cardiovascular surgery intensive care units
* To answer the survey questions

Exclusion Criteria:

* To Working or worked in cardiovascular surgery intensive care unit and but not answering questionnaire questions

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: physiotherapists working in cardiovascular intensive care
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Delivery of surveys | 1 month
  Questionnaire questions will be sent to physiotherapists via mail or telephone
Evaluation of survey results | 4 months
  Statistical evaluation and interpretation of survey results

CONTACTS AND LOCATIONS:
Overall Officials: Halime Sinem Barutçu, Principal Investigator; Hatun İlkatmış İnce, Principal Investigator; Füsun Güzelmeriç, Study Director
Locations (1):
- Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
communicating with physiotherapists mail sending evaluation of answers interpretation of results

REFERENCES:
- [Background] Westerdahl E, Olsen MF. Chest physiotherapy and breathing exercises for cardiac surgery patients in Sweden--a national survey of practice. Monaldi Arch Chest Dis. 2011 Jun;75(2):112-9. doi: 10.4081/monaldi.2011.223. PMID 21932695
- [Background] Reeve J, Denehy L, Stiller K. The physiotherapy management of patients undergoing thoracic surgery: a survey of current practice in Australia and New Zealand. Physiother Res Int. 2007 Jun;12(2):59-71. doi: 10.1002/pri.354. PMID 17536644
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/20738852
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/17536644